CLINICAL TRIAL: NCT03122210
Title: Comparaison of 2 SpO2 Level Measured by Pulse Oxymetry in Complications of Acute Coronary Syndrome.
Acronym: FreeO2 SCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, François Lellouche, Principal investigator, Laval University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20502
Record Dates: First submitted 2017-04-18; First posted 2017-04-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-12

CONDITIONS: Infarction, Myocardial
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Other): In this group, the nursing staff administed oxygen supply if necessary with the usual pratice in care unit for 24 hours after myocard infarction. In this group the SpO2 was recorded any time with FreeO2 device - recording mode.
  Interventions: Device: Automated oxygen administration
- FreeO2 with SpO2 target = 92% (Other): In this group oxygen flow was automatically adjusted with the FreeO2 device (automatic titration of oxygen flow) to achived SpO2 target set by clinicial for 24 hours after myocard infarction. In this group, the SpO2 target was set at 92%.
  Interventions: Device: Automated oxygen administration
- FreeO2 with SpO2 target =97% (Other): In this group oxygen flow was automatically adjusted with the FreeO2 device (automatic titration of oxygen flow) to achived SpO2 target set by clinicial for 24 hours after myocard infarction. In this group, the SpO2 target was set at 97%.
  Interventions: Device: Automated oxygen administration

INTERVENTIONS:
Device: Automated oxygen administration — In the control group, usual oxygen administration and titration is planned
  Other Names: Usual oxygen administration

SUMMARY:
During acute coronary syndrome, the American College of Cardiology and the American Heart Association recommend oxygen delivery to patients with less than 90% oxygen saturation. Oxygen therapy in these patients for a duration of at least 6 hours, but also stipulates that it is reasonable to administer oxygen to all acute coronary syndrome patients during the first six hours following the presentation. Hyperoxia also has well-established risks.

Our research hypotheses are:

(I) that current practices tend to use high oxygen flows resulting in high SpO2 levels during acute coronary syndrome.

(II) there is a high rate of desaturation in patients with acute coronary syndrome and an automatic adaptation of oxygen flows may reduce this frequency.

(III) that excessive oxygenation targets have no advantage. Our hypothesis is that maintaining a SpO2 of 90 to 94% is at least equivalent when compared to higher saturation objectives (SpO2 of 94 to 100%) with regard to the occurrence of complications in the patient in acute coronary syndrome . We will use two SpO2 targets with the FreeO2 system, 92 and 97%.

DETAILED DESCRIPTION:
Hypoxemia is a common problem encountered during acute coronary syndrome. During acute coronary syndrome, the American College of Cardiology and the American Heart Association recommend oxygen delivery to patients with less than 90% oxygen saturation. Oxygen therapy in these patients for a duration of at least 6 hours , but also stipulates that it is reasonable to administer oxygen to all acute coronary syndrome patients during the first six hours Following the presentation. However, the studies underlying these guidelines are few and far between, most of them having been done more than forty years ago.

Hyperoxia also has well-established risks.

Our research hypotheses are:

(I) that current practices tend to use high oxygen flows resulting in high SpO2 levels during acute coronary syndrome.

(II) there is a high rate of desaturation in patients with acute coronary syndrome and an automatic adaptation of oxygen flows may reduce this frequency. This will be our primary endpoint and will be tested with the use of the automated oxygen delivery system.

(III) that excessive oxygenation targets have no advantage. Our hypothesis is that maintaining a SpO2 of 90 to 94% is at least equivalent when compared to higher saturation objectives (SpO2 of 94 to 100%) with regard to the occurrence of complications in the patient in acute coronary syndrome . We will use two SpO2 targets with the FreeO2 system, 92 and 97%.

ELIGIBILITY:
Inclusion Criteria:

* Patients should have a proven diagnosis of acute high risk coronary syndrome as defined by the American Heart Association:
* myocardial infarction with or without ST segment elevation: Ischemic changes in the electrocardiogram and positive cardiac biomarkers.
* or Unstable angina: Typical or atypical cardiac symptoms, Ischemic electrocardiographic changes, Normal cardiac biomarkers.

Exclusion Criteria:

* inclusion in another study refusing co-enrollment
* chronic obstructive pulmonary disease with CO2 retention
* sleep apnea-hypopnea syndrome with CPAP
* traumatic brain injury
* pregnancy
* Age <18 years
* Mechanical invasive or non-invasive ventilation
* patient needing more than 5 lpm of oxygen to have SpO2 > 95%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01-05 (Actual); Primary Completion 2013-08-08 (Actual); Study Completion 2017-04-13 (Actual)

PRIMARY OUTCOMES:
The frequency of significant desaturations (SpO2 <90% for at least 30 seconds) | 24 hours

SECONDARY OUTCOMES:
Significant rhythm disorders, ischemic events | 24 hours
The percentage of time spent in the target SpO2 area in the second and third groups, defined as SpO2 +/- 2% of the targeted SpO2 (range 90-94% for group 92% and range 95-99% for group 97%) | 24 hours

IPD SHARING:
Plan to Share IPD: Undecided